CLINICAL TRIAL: NCT01104506
Title: Elaboration of a Pre-surgery Mapping Protocol of Primary Motor Cortex, Prior to an Implementation of a Stimulation of Primary Motor Cortex for Patients With Deafferentiation of Brachial Plexus Pain
Acronym: CCPB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Anne OMNES, Nantes University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BRD 10/2-A; 2010-A00141-38 (Other: Afssaps)
Record Dates: First submitted 2010-04-08; First posted 2010-04-15 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-04

CONDITIONS: Painful Avulsion of Brachial Plexus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Painless plexus (Active Comparator): Patient with a painless avulsion of brachial plexus
  Interventions: Procedure: fMRI; Procedure: mTMS
- Healthy (Active Comparator): Healthy volunteers
  Interventions: Procedure: fMRI; Procedure: mTMS
- Painful plexus (Experimental): Patient with a painful avulsion of brachial plexus
  Interventions: Procedure: fMRI; Procedure: mTMS

INTERVENTIONS:
Procedure: fMRI
Procedure: mTMS

SUMMARY:
In the context of an insufficiency of clinical results for cortical stimulation in treatment of brachial plexus post-avulsion pains, one of the possibility for failure is the bad pre-surgery mapping of the area to stimulated bu the usual methods (PEM et fMRI). This purpose of this study is to realise a precise mapping of the primary motor cortex post brachial plexus avulsion.

The principal endpoints is to identify and test the reliability of a muscular marker for which the cortical representation is localized immediately next to the superior member area. Several muscles of cephalic, cervical and chest area will be investigate.

The methods used will be mono-shock transcranial magnetic stimulation (mTMS) and functional MRI.

Concerning mTMS, several methods will be tested: best position on the scalp, realisation of outputs maps with extreme points average method, with mass center method.

Concerning fMRI studies, the above paradigms will be checked: imaginary movements of hand, blow up and down abdomen, eyes winking.

Statistical tests will confirm the best muscle candidate and will permit to evaluate the reliability of the method.

ELIGIBILITY:
Inclusion Criteria:

* For all groups: informed consent, social insurance
* For group 1 "painful BPA": consulting to the Nantes'UH for pain of BPA, EVA≥4, neurological deficiency partial or total
* For group 2 "painless BPA": EVA<4, neurological deficiency partial or total, matching with group 1 on the neurological deficiency
* For group 3 "Healthy": matching with group 1 on age ±10 years

Exclusion Criteria:

* No informed consent
* Medical history of epilepsy
* Pregnant women
* Contra-indication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Identify the 2 muscles (lateral and medial) lining the representation of superior member according to Penfield's homunculus.
  Spatial coordinates (xyz): calculation of the center of gravity of cortical surface suggestive of a specific muscle, using data acquired during each session.

SECONDARY OUTCOMES:
Evaluation of primary outcome depending on cortical center
  Calculation of cortical center evoking the maximal PEM
Evaluation of primary outcome depending on the center of cortical area
  Calculation of the center of the cortical area suggestive of a precised muscle
Evaluation of primary outcome depending on cortical surface
  Calculation of cortical surface suggestive of a precised muscle
Pain intensity
  Pain intensity by using an visual analogic scale
Ghost sensations intensity
  Ghost sensations intensity by a questionnaire
Amplitude of PEM
  calculation of the amplitude of PEM for a precised muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes UH, Nantes, France